CLINICAL TRIAL: NCT05426642
Title: Development and Evaluation of KaSEH Video to Increase Women's Knowledge and Motivation Regarding Cervical Cancer and Its Screening.
Brief Title: The Effect of E-health Video Towards Enhancing Cervical Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: FF-2021-499
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receive the e-health video and brochure as the intervention
  Interventions: Other: E-health Video KaSEH; Other: Brochure
- Control group (Other): Receive brochure as the intervention
  Interventions: Other: Brochure

INTERVENTIONS:
Other: E-health Video KaSEH — The e-health video KaSEH is produce based on Protection Motivation Theory to enhance women's motivation towards cervical cancer screening.
  Arms: Intervention group
Other: Brochure — The brochure contain the information regarding cervical cancer and its screening

SUMMARY:
The aim of this quasi-experimental study is to evaluate the women's motivation related to cervical cancer screening. The experiment group will receive the e-health video KaSEH and brochure as the intervention. Where as, the control group will receive brochure as the intervention. There is three phase of evaluation which are pre-intervention, intra-intervention and post-intervention. The evaluation will be assess using the self-administered questionnaire based on Protection Motivation Theory. The estimated duration of this quasi-experiment is six month.

ELIGIBILITY:
Inclusion Criteria:

* Women who have never undergone cervical cancer screening.

Exclusion Criteria:

* Women who have been diagnosed or are cervical cancer patients
* Women who have been diagnosed with any cancer of the gynecological system such as cancer of the vulva, vagina, uterus, fallopian tubes and ovaries.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Motivation level | 3 month
  The score of motivation level measured by means (standard deviation) using The Malay-Protection Motivation Theory scale for cervical cancer screening as measurement tool.
Practice | 3 month
  Measured by yes (uptake of cervical cancer screening) and no (did not perform screening).